CLINICAL TRIAL: NCT00192322
Title: A Randomized, Partially-Blinded, Placebo-Controlled Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine, Trivalent,Types A & B, Live Cold Adapted (CAIV-T) in Healthy Children Aged 6 to Less Than 36 Months
Brief Title: Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine (CAIV-T) in Healthy Children
Acronym: CAIVT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Raburn Mallory, MD/ Sr Dir Clinical Development, MedImmune
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D153-P002
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CAIV-T 10^5 (Experimental): a single intranasal 0.2 mL dose of liquid CAIV-T 10^5 (approximately 0.1 mL into each nostril)
  Interventions: Biological: CAIVT 10^5
- CAIVT 10^7 (Experimental): A single intranasal 0.2 mL dose of liquid CAIV-T 10^7 (approximately 0.1 mL into each nostril)
  Interventions: Biological: CAIV-T 10^7
- Placebo (Placebo Comparator): A single intranasal 0.2 mL dose of placebo
  Interventions: Biological: Placebo
- Trivalent inactivated vaccine (TIV) (Active Comparator): A single intramuscular injection of commercially available vaccine
  Interventions: Biological: TIV

INTERVENTIONS:
Biological: CAIV-T 10^7 — a single intranasal 0.2 mL dose of liquid CAIV-T 107 (approximately 0.1 mL into each nostril)
  Arms: CAIVT 10^7
Biological: CAIVT 10^5 — a single intranasal 0.2 mL dose of CAIV-T <10^5
  Arms: CAIV-T 10^5
Biological: Placebo — a single intranasal 0.2 mL dose of placebo
  Arms: Placebo
Biological: TIV — commercially available TIV injected intramuscularly
  Arms: Trivalent inactivated vaccine (TIV)

SUMMARY:
To perform a variety of assays on blood, nasal washes, and cells obtained from healthy children for the purposes of further investigation of immune responses generated by influenza virus vaccine, trivalent, types A and B, live, cold-adapted (liquid CAIV-T; Wyeth Lederle Vaccines, Marietta, PA).

• To assess nasal swab specimens to detect vaccine virus shedding.

DETAILED DESCRIPTION:
This was a phase II, prospective, randomized, partially-blinded, placebo-controlled, outpatient study conducted at multiple sites throughout the US in healthy children aged 6 months to less than 36 months. Parents/guardians of subjects were asked to read and sign the informed consent before any study-related procedures were performed. Subjects at each study site were sequentially assigned to 1 of 2 separate blood sample groups referred to as "cellular immunity" or "antibody secreting cell". Subjects within each blood sample group were then randomized 1:1:1:1 to receive a single intranasal dose of CAIV-T 10^7 FFU per dose, CAIV-T 10^5 FFU per dose, placebo or a commercially-available injectable trivalent influenza vaccine (TIV).

ELIGIBILITY:
Inclusion Criteria:

* children at least 6 months of age and less than 36 months of age at the time of enrollment, and in good health as determined by medical history, physical examination and clinical judgement;
* whose parent/legal guardian has provided written informed consent after the nature of the study has been explained;
* who, along with their parent or guardian, will be available for the one month duration of the trial (from enrollment to study completion);

Exclusion Criteria:

* whose parents or guardians are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids, or cytotoxic agents (see Section 4.2.2);
* have an immunosuppressed or an immunocompromised individual living in the same household;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine, placebo or TIV;
* who, at anytime prior to study enrollment, receives any influenza vaccine (commercial or investigational);
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results.

Note: A pregnant household member is not considered a contraindication to enrollment.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2001-09; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Measurement of influenza-specific immune response following receipt of CAIV-T. | Day 0 and Day 27
  The immune responses were evaluated by hemagglutination inhibition assay (HAI) on serum samples.

SECONDARY OUTCOMES:
Vaccine virus shedding | Days 2, 6, and 13
  The number of subjects who shed influenza virus vaccine subtypes following vaccination.
Measurement of influenza-specific immune response following receipt of CAIVT. | Day 0 and Day 27
  The immune responses were evaluated by mucosal IgA ELISA on nasal wash samples.
Measurement of influenza-specific immune responses following receipt of CAIVT | Day 0, Day 6, and Day 13
  The immune responses were evaluated by assays of cellular immunity (IFN-gamma ELISPOT) and assays that measured the number of antibody secreting cells (B-cell ELISPOT).
Assess the safety and tolerability of CAIV-T vaccine in healthy children. | Day 0-27
  Adverse events and serious adverse events were collect from Day 0 till the end of the study Day 27.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Principal Investigator — MedImmune LLC
Locations (2):
- United States (2):
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Division of Allergy Immunology and Infectious Disease, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Mendelman PM, Rappaport R, Cho I, Block S, Gruber W, August M, Dawson D, Cordova J, Kemble G, Mahmood K, Palladino G, Lee MS, Razmpour A, Stoddard J, Forrest BD. Live attenuated influenza vaccine induces cross-reactive antibody responses in children against an a/Fujian/411/2002-like H3N2 antigenic variant strain. Pediatr Infect Dis J. 2004 Nov;23(11):1053-5. doi: 10.1097/01.inf.0000143643.44463.b1. PMID 15545863